CLINICAL TRIAL: NCT00825708
Title: Evaluation of the Effect of rTMS on Attention in Adults Diagnosed With ADHD
Brief Title: Evaluation of the Effect of rTMS on Attention in Adults Diagnosed With Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Yuval Bloch, shalvataMHC
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SH20107; SH20107
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS (Active Comparator): rTMS session
  Interventions: Device: rTMS
- SHAM (Sham Comparator): sham session
  Interventions: Device: shamTMS

INTERVENTIONS:
Device: rTMS — 42 2 sec trains of 20HZ rTMS in 100% MT
  Arms: rTMS
Device: shamTMS — sham TMS session
  Arms: SHAM

SUMMARY:
The aim of the study is to evaluate the immediate effect of rTMS on attention in adults diagnosed with ADHD. the design is a double blind sham controlled crossover study.

DETAILED DESCRIPTION:
The subjects were randomly assigned to two groups. group 1 starts with the real rTMS session followed within one week with a sham session. group 2 starts with a sham session and within one week recieve a real session. the subjects go through a neurocognitive evaluation before and after rTMS sessions and a clinical evaluation questionnaire modified for attention.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* diagnosis of ADHD according to DSM IV criteria

Exclusion Criteria:

* other axis I diagnosis
* risk factors for seizure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
PANNAS questionnaire modified for attention | within one hour of the rTMS session

SECONDARY OUTCOMES:
the CANTAB neurocognitive battery | within 2 hours of the stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata MHC, cognitive and emotion lab, Hod HaSharon, Israel

REFERENCES:
- [Derived] Bloch Y, Harel EV, Aviram S, Govezensky J, Ratzoni G, Levkovitz Y. Positive effects of repetitive transcranial magnetic stimulation on attention in ADHD Subjects: a randomized controlled pilot study. World J Biol Psychiatry. 2010 Aug;11(5):755-8. doi: 10.3109/15622975.2010.484466. PMID 20521875